Version 15-Dic 2020. Informed consent form. *Risk factors to develop chronic postsurgical pediatric pain*.





## CHRONIC POSTSURGICAL PEDIATRIC PAIN.

**TITLE:** RISK FACTORS TO DEVELOP CHRONIC POSTSURGICAL PEDIATRIC PAIN

**INVESTIGATOR PRINCIPAL:** GUILLERMO CENIZA-BORDALLO

**PROJECT ENTITIES:** COMPLUTENSE UNIVERSITY OF MADRID & 12 OCTUBRE PEDIATRIC HOSPITAL.

**NUMBER OF IDENTIFIACTION:** 26/618

**DATE:** 15<sup>TH</sup> December 2020.

Version 15-Dic 2020. Informed consent form. Risk factors to develop chronic postsurgical pediatric pain.





SI/NO

## **INFORMED CONSENT FORM**

Research Project title: RISK FACTORS TO DEVELOP CHRONIC POSTSURGICAL PEDIATRIC PAIN

## The legal guardian should read and answer the questions paying attention

Have you reded all information with this project?

| • | Had you the opportunity to ask all questions about project? | SI / NO |
|---|---|---|
| • | Have you received satisfactoriness' answers? | SI / NO |
| • | ve you have understood that your child is free to abandon this project without this | |
| | decision being able to cause you any harm? | SI/NO |
| • | Anytime? | SI / NO |
| • | Without no reasons? | SI / NO |
| • | Are you agree with you child participation in this project? | SI / NO |
| • | Will you receive any economic compensation for your child participation in this | eceive any economic compensation for your child participation in this Project? |
| | | SI / NO |

Do you authorize the participation in the project of the person for whom you are responsible? (By signing the consent form, you agree to comply with the study procedures that have been exposed to you).

SI / NO

Version 15-Dic 2020. Informed consent form. Risk factors to develop chronic postsurgical pediatric pain.

| Name and surname of the volunteer's legal guardian: |
|---------------------------------------------------------------------|
| Firm of volunteer's legal guardian: |
| Date |
| Phone number of volunteers' legal guardian: |
| Are you agree with your participation in this project? (+ 12 years) |
| Name and surname of volunteer: |
| Firm of volunter: |
| Date |